CLINICAL TRIAL: NCT04579016
Title: Pragmatic Lifestyle Pregnancy and Post Pregnancy Intervention for Overweight Women With Gestational Diabetes Mellitus: a Randomised Controlled Clinical Trial (PAIGE2)
Brief Title: Pragmatic Lifestyle Pregnancy and Post Pregnancy Intervention for Overweight Women With Gestational Diabetes Mellitus
Acronym: PAIGE2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Belfast Health and Social Care Trust (Other)
Collaborators: Northern Health and Social Care Trust (Other Government); South Eastern Health and Social Care Trust (Other); Interreg (Other); Our Lady of Lourdes Hospital, Drogheda (Other Government); Sligo General Hospital (Other); Letterkenny University Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 18/NI/0228
Record Dates: First submitted 2020-10-01; First posted 2020-10-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Weight Loss; Gestational Diabetes
MeSH Terms: conditions — Weight Loss; Diabetes, Gestational | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care (Active Comparator): Standard care
  Interventions: Other: Standard care
- PAIGE2 intervention (Experimental): One hour education session during pregnancy. Postnatally provision of activity tracker, 3/6 month referral to a commercial weight management organization, text and phone support.
  Interventions: Other: PAIGE2 lifestyle intervention

INTERVENTIONS:
Other: PAIGE2 lifestyle intervention — Education session during pregnancy. provision of fitness tracker, referral to commercial weight management organization, text and phone support
  Arms: PAIGE2 intervention
Other: Standard care — Care routinely provided to all pregnant women diagnosed with GDM
  Arms: Standard care

SUMMARY:
This study is designed to determine if a postnatal lifestyle intervention will lead to weight reduction over a 12 month period post-delivery in women who have been diagnosed with gestational diabetes mellitus and who have a BMI greater that 25 compared to women who receive routine care.

DETAILED DESCRIPTION:
Diabetes during pregnancy (Gestational Diabetes Mellitus (GDM) is defined as high blood sugars during pregnancy and it is becoming increasingly common which affects around 18% of pregnant women. GDM is usually diagnosed by an oral glucose tolerance test around 28 weeks gestation. Women with previous GDM have a 50% risk of developing it again in any future pregnancy, and are 7 times more likely to develop type 2 diabetes within the future compared to women without GDM.

There is evidence that lifestyle changes (diet and physical activity), can reduce the development of type 2 diabetes in people at high risk, such as women with previous GDM. The postnatal period (shortly after pregnancy) is an ideal time for women to make these changes to help prevent weight gain between pregnancies and generally reduce their risk of future type 2 diabetes. This study is designed to determine if a postnatal lifestyle intervention will lead to weight reduction over a 12 month period post-delivery.

Women who have been diagnosed with diabetes during pregnancy (GDM) and had a body mass index (BMI) >25 kg/m2 at the start of pregnancy, will be invited to take part in the study.

During their routine appointment at 32-36 weeks gestation women will be randomly allocated either to the intervention program or control group.

Women in the intervention group, will receive a 1-hour educational session during their routine diabetes antenatal clinic visit. In addition, they will be offered an activity tracker (following consent) to help monitor their daily step count and physical activity.

Women in both the intervention and control groups will have a fasting glucose blood sample taken the morning after delivery. Those women with normal or borderline fasting glucose levels are eligible to remain in the study, but those with type 2 diabetes will be excluded and referred to their local diabetes team.

At 6-8 weeks postnatally, both groups will complete some questionnaires, give a blood sample, have weight and blood pressure measurements recorded. Women will be offered free referral to a commercial weight management organization for 12 weeks, with a possible extension for another 12 weeks). Over the 12 months of the study, the PAIGE2 team will contact participants intermittently by text and telephone to encourage them to eat healthily and increase their physical activity. If the participants' partner is also willing to take part, the partner will be sent an activity tracker to monitor physical activity and the research team will keep in intermittent contact with the partner by text and telephone during the study.

Women allocated to the control group will be offered a free 12-week referral to a commercial weight management organization at the end of the study.

Both groups will be asked to attend 2 further study visits at 6 and 12 months after delivery. This will involve completion of some questionnaires, a blood test, weight and blood pressure measurements.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 18 years of age or older,
2. Women with a booking BMI ≥ 25 kg/m2 at <14 weeks gestation
3. GDM has been diagnosed in their current pregnancy.
4. Women will only continue to be included in the study if their fasting plasma glucose the morning after delivery indicates normality or impaired fasting plasma glucose outside of pregnancy (i.e.<7 mmol/l).
5. Women with a history of GDM directly preceding the current pregnancy, and who were given lifestyle advice and were performing self-monitoring of blood glucose from early pregnancy, will also be included if capillary glucose monitoring exceeds target values (fasting ≥ 5.3 mmol/l (95 mg/dl), 1h postprandial plasma glucose ≥ 7.8 mmol/l (140 mg/dl) thus negating the need for an OGTT.

   -

   Exclusion Criteria:

   Pregnancy in which an anomaly has been detected on the 20-week fetal anomaly scan.

b.) History of diabetes outside of pregnancy or FPG ≥7 mmol/l the morning after delivery.

c.) History of heart, liver or chronic renal disease. d.) Medications that adversely affect glucose tolerance (e.g. steroids). e.) Inability to participate in moderate physical activity outside of pregnancy.

f.) Moderate/severe depressive illness or excess alcohol consumption. g.) Inability to understand adequately verbal explanations or written information in English, or special communication needs.

h.) Women who are planning another pregnancy within the next 12 months following delivery.

i.) Exclusion criteria for early post-partum glucose testing will include massive postpartum hemorrhage, steroid treatment prior to delivery or patient refusal.

* If a woman requests an earlier discharge that does not allow time for the FPG test, she will be offered an appointment to return to the maternity unit within four weeks of birth for retesting.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-01-13 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Weight loss | Change from baseline to 12 months postpartum
  Weight loss

SECONDARY OUTCOMES:
Fasting glucose | Change from baseline to 12 months postpartum
  Fasting glucose
Waist circumference | Change from baseline to 12 months postpartum
  Waist circumference
Step counts (intervention group only) | Change from baseline to 12 months postpartum
  Number of steps taken
Questionnaire data pertaining to physical activity, General Health and Well Being, Motivation to change and Risk Perception Survey for Developing Diabetes | Change from baseline to 12 months postpartum
  Questionnaire data

CONTACTS AND LOCATIONS:
Overall Officials: David McCance, Principal Investigator — Belfast Health and Social Care Trust
Locations (1):
- Royal Victoria Hospital, Belfast, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McAuley E, Fleck O, Cassidy L, Kemp BJ, Cupples G, Kelly B, Creighton RM, Graham U, Wallace H, Patterson CC, McCance DR. A pragmatic lifestyle intervention for overweight and obese women with gestational diabetes mellitus (PAIGE2): A parallel arm, multicenter randomized controlled trial study protocol. Front Clin Diabetes Healthc. 2023 Mar 24;4:1118509. doi: 10.3389/fcdhc.2023.1118509. eCollection 2023. PMID 37034478